CLINICAL TRIAL: NCT05749159
Title: Comparison of New pHysIotherapy With Alternative Therapy for Clinical outComes in Patients With hiccUP: Rationale and Design of a Randomized Clinical Trail
Brief Title: New Physitherapy or Alternative Therapy for Hiccup
Acronym: HICCUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0115
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Hiccup
Keywords: hiccup
MeSH Terms: conditions — Hiccup | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiotherapy (Experimental): New physical therapy: a disposable cup (soft cup) to take 1/3 cup of room temperature water and place it on a table. The patient takes a sitting or standing position. The middle finger of both hands press tightly against the nose to seal the nasal cavity. At the same time, press the ear screen with both hands to close the ear canal. After that, bite the cup with teeth (hands do not touch the cup), and drink up 1-2 mouthfuls of water.
  Interventions: Behavioral: physiotherapy
- alternative therapy (Placebo Comparator): Alternative therapy: including routine physical therapy such as suffocation and drinking cold water, as well as drug therapy such as metoclopramide and Mianna.
  Interventions: Behavioral: physiotherapy

INTERVENTIONS:
Behavioral: physiotherapy — New physical therapy: a disposable cup (soft cup) to take 1/3 cup of room temperature water and place it on a table. The patient takes a sitting or standing position. The middle finger of both hands press tightly against the nose to seal the nasal cavity. At the same time, press the ear screen with both hands to close the ear canal. After that, bite the cup with teeth (hands do not touch the cup), and drink up 1-2 mouthfuls of water.

SUMMARY:
Hiccup is a common symptom, and it is currently believed that hiccups result from diaphragmatic spasm, with onset ranging from minutes to days. Some patients may terminate on their own, or by ways such as gasping. For some patients with duration longer than 1 day, even longer than 2 days, medications may be needed, mainly: metoclopramide, eperisone hydrochloride tablets, etc. Acupuncture is also effective for some patients. Surgical treatment may be required for some clinically intractable hiccups. However, for the above interventions or treatment means, the current efficacy still needs to be improved.

In the previous clinical experience, we create a new physical clinic protocol which could terminate the hiccup symptom onset instantaneously without adding extra cost to the patient, and the physiotherapy method was convenient and effective. To further validate the superiority, safety of this novel physical therapy regimen, we designed a randomised controlled, prospective, single centre clinical study aimed at comparing the efficacy and safety of the novel physical therapy with conventional pharmacotherapy in patients with hiccups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to swallow water

Exclusion Criteria:

* Allergy or contraindication to the following drugs: metoclopramide et al
* Severe choking on water and difficulty swallowing were present
* Impaired consciousness and inability to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of termination of hiccup in 30 seconds | 1 year
  the rate of termination of hiccup in 30 seconds
the time course from the start of therapy to the end of hicuup | 1 year
  the time course from the start of therapy to the end of hicuup

CONTACTS AND LOCATIONS:
Overall Officials: Shen Jian, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No